CLINICAL TRIAL: NCT05140954
Title: Safety and Pharmacokinetics of TAF-FTC Pre-exposure Prophylaxis in Kenyan Cisgender Women
Brief Title: The Women TAF-FTC Benchmark Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Kenya Medical Research Institute (Other); University of Colorado, Denver (Other); Gilead Sciences (Industry)
Responsible Party: Principal Investigator, Kenneth K Mugwanya, Assistant Professor, University of Washington
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00014075; CO-US-412-6203 (Other Grant/Funding Number: Gilead Sciences)
Record Dates: First submitted 2021-11-18; First posted 2021-12-02 (Actual); Results first posted 2025-10-27 (Actual); Last update posted 2025-10-27 (Actual); Status verified 2025-09

CONDITIONS: HIV Infections
Keywords: Pre-exposure Prophylaxis; HIV; Kenya; Descovy
MeSH Terms: conditions — HIV Infections | interventions — Racivir; emtricitabine tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Perfect Adherence (Experimental): Cisgender women will receive a single tablet of coformulated 25 mg TAF/ 200mg FTC once daily (7 doses per week).
  Interventions: Drug: co-formulated 25mg TAF/ 200mg FTC
- Moderate Adherence (Experimental): Cisgender women will receive a single tablet of coformulated 25 mg TAF/ 200mg FTC 4 times per week
  Interventions: Drug: co-formulated 25mg TAF/ 200mg FTC
- Poor Adherence (Experimental): Cisgender women will receive a single tablet of coformulated 25 mg TAF/ 200mg FTC twice per week
  Interventions: Drug: co-formulated 25mg TAF/ 200mg FTC

INTERVENTIONS:
Drug: co-formulated 25mg TAF/ 200mg FTC — Participants will be randomized into 1 of 3 groups to receive a controlled number of doses of a single tablet of co-formulated 25 mg TAF/ 200mg FTC
  Other Names: Descovy

SUMMARY:
The study seeks to assess the safety of and define blood and tissue benchmark concentrations of tenofovir diphosphate (TFV-DP) and emtricitabine triphosphate (FTC-TP) in cisgender women using directly observed oral pre-exposure prophylaxis (PrEP) therapy with tenofovir alafenamide-emtricitabine (TAF-FTC). Cisgender women will be randomly assigned to receive varying frequencies of weekly PrEP doses and followed for up to 18 weeks.These data will help accurate interpretation of efficacy results obtained in HIV prevention trials and programs in cisgender women.

DETAILED DESCRIPTION:
This is an open-label, randomized, three-arm, directly observed therapy (DOT), pharmacokinetics study. HIV-uninfected non-pregnant cisgender women at low risk for HIV acquisition will be randomly assigned to 1 of 3 dosing frequencies of DOT with tenofovir alafenamide-emtricitabine (TAF-FTC) oral PrEP, to help differentiate poor and moderate from perfect adherence. The primary objectives of the study are:

1. To describe the safety of TAF-FTC-based PrEP in HIV-uninfected cisgender women.
2. To define expected blood concentrations and dose-proportionality specific to cisgender women for tenofovir-diphosphate (TFV-DP) in dried blood spots (DBS) and peripheral blood mononuclear cells (PBMCs) using directly observed therapy of TAF-FTC at 2, 4, and 7 doses per week, representing poor, moderate, and perfect adherence, respectively.
3. To establish a model to predict adherence rate to TAF-FTC by level of TFV-DP in DBS for cisgender women. HIV-uninfected non-pregnant cisgender women will be randomly assigned to 1 of 3 dosing frequencies of directly observed therapy of TAF-FTC oral PrEP: 2, 4, or 7 doses/week to differentiate poor and moderate from perfect adherence.

The study will be the first to define TAF-FTC-based PrEP adherence-blood concentration thresholds for African cisgender women, a priority population for HIV prevention. The findings will guide accurate interpretation of safety, adherence, and efficacy of planned or ongoing HIV prevention trials in African women.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤30 years old
* Willing to undergo urine pregnancy tests
* Has understood the information provided and has provided written informed consent before any study-related procedures are performed.
* HIV uninfected based on negative HIV rapid tests, according to Kenyan national algorithm
* Normal renal function (estimated glomerular filtration rate >60 mL/min)
* Hepatitis B surface Ag negative
* No active clinically significant medical or psychiatric conditions that, in the opinion of the investigators, would interfere with study participation
* Lack of severe anemia (Hemoglobin >10 g/dL)
* Willing to use DOT and come to clinic frequently for DOT PrEP for at least 10 weeks
* Willing to have home visits for follow up
* Has access to an active smartphone to allow off-site observation of dosing if unable to come to the clinic or as determined by the study staff, the participant resides in close location to clinic to permit home visit if unable to come to the clinic. i.e., potential participants without a smartphone may be enrolled in the study if investigator determines that the participant resides within reasonable distance from the clinic that would permit home visit id the participant misses their visit.
* Intention to stay within the study site's catchment area for at least 10 weeks.
* Resides or works in catchment area with high speed internet coverage to permit video streaming
* Not pregnant or breast feeding
* Willing to use effective contraception during the study period.
* At low risk for HIV. In Kenya, national guidelines define substantial risk for HIV and recommend PrEP be an option for individuals reporting: partner of HIV-infected person not on ART or on ART for <6 months, >1 partner of unknown status, transactional sex, recent STI, recurrent PEP use, inconsistent condom use, or injection drug use. So, non-pregnant cisgender women reporting any of these factors will not be eligible for the study but will be linked for PrEP at clinic of choice including at Thika Site itself.
* Willing to be randomized to non-daily PrEP and come to clinic frequently for DOT PrEP
* Willingness and ability to be abstinent for at least 7 days after each vaginal biopsy visit.

Exclusion Criteria:

* Inability to give informed consent
* Positive screening HIV+ as determined by standard rapid serologic assays or suspected acute HIV infection in the opinion of the clinician. (example signs and symptoms of acute HIV infection include combinations of fever, headache, fatigue, arthralgia, vomiting, myalgia, diarrhea, pharyngitis, rash, night sweats, and adenopathy cervical or inguinal)
* Positive HBV surface antigen test at screening
* Calculated creatinine clearance <60 ml/min.
* Any laboratory value or uncontrolled medical conditions that, in the opinion of the investigators, would interfere with the study conditions such as, heart disease and/or cancer.
* Prohibited concomitant medications are: investigational agents (within 30 days of enrollment), aminoglycosides, ganciclovir/valganciclovir, chronic high-dose acyclovir/valacyclovir (>800mg acyclovir or >500mg valacyclovir for >7 days), cyclosporine, amphotericin B, foscarnet, and cidofovir, and products with same or similar active ingredients as the study medications including TAF®, TRUVADA®, ATRIPLA®, COMPLERA®, EMTRIVA®, VIREAD®; or drugs containing lamivudine or adefovir, which are close analogs of FTC and tenofovir, respectively.
* Current or past use of PrEP (pre-exposure prophylaxis)
* Not willing to have home visits
* Pregnancy or plan to become pregnant in the next 6 months or unwillingness to use birth control
* Current breastfeeding
* High risk of HIV infection (for example: sexually active with an HIV infected partner; engages in condomless intercourse with HIV-infected partners or partner of unknown status during the study; females who exchange sex for money, shelter, or gifts; active injection drug use or during the last 12 months; newly diagnosed sexually transmitted infections in last 6 months.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2023-03-28 (Actual); Primary Completion 2023-12-19 (Actual); Study Completion 2023-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth K Mugwanya, MBChB, MS, PhD, Principal Investigator — University of Washington; Peter L Anderson, PharmD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Kenya Medical Research Institute - Partners in Health Research and Development, Thika, Kenya

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Seventy-one women were screened for study participation starting 28 March 2023 to 11 September 2023 at the Kenya Medical Research Institute, Center for Clinical Research, Thika site in Kenya. The Of these, 54 healthy volunteer women ages 18-30 at low risk of HIV acquisition were enrolled into the study and randomized. The first participant was randomized on 10 April 2023.
Period: Overall Study
Arm/Group | Poor Adherence | Moderate Adherence | Perfect Adherence
Started | 18 | 18 | 18
Completed | 16 | 17 | 18
Not Completed | 2 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Poor Adherence | Moderate Adherence | Perfect Adherence | Total
Number analyzed (Participants) | 18 | 18 | 18 | 54
Age, Customized [Median (Inter-Quartile Range); unit: years]
  Median age | 22 [20.5 to 24] | 24.5 [22 to 28] | 23 [21 to 24] | 23 [21 to 25]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 18 | 18 | 54
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Kenya | 18 | 18 | 18 | 54

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Adverse Events
Description: The frequency of graded adverse events by arm, including emergent HIV infection during the study period.
Time Frame: Assessed through the 10 week DOT dosing period
Measure: Number; unit: Number of adverse events
Arm/Group | Poor Adherence | Moderate Adherence | Perfect Adherence
Number analyzed (Participants) | 18 | 18 | 18
Number of adverse events
  Grade 1 adverse events | 69 | 60 | 62
  Grade 2 adverse events | 1 | 1 | 0
  Grade 3 or higher adverse events | 0 | 0 | 0
  Emergent HIV infection | 0 | 0 | 0

2. Primary Outcome: Concentrations of Tenofovir Disphosphate (TFV-DP) and Emtricitabine Triphosphate (FTC-TP) Measured at Ten Weeks in Dried Blood Spots (DBS)
Description: TFV-DP and FTC-TP concentrations observed in dried blood spots (DBS) after ten weeks of directly observed therapy with TAF-FTC oral PrEP, in women randomized to receive 2, 4, or 7 doses per week, representing poor, moderate, or perfect adherence, respectively.
Time Frame: Assessed at week 10
Measure: Median (Inter-Quartile Range); unit: fmol/punches
Arm/Group | Poor Adherence | Moderate Adherence | Perfect Adherence
Number analyzed (Participants) | 16 | 17 | 18
fmol/punches
  Observed TFV-DP concentrations | 432 [407 to 504] | 1214 [930 to 1377] | 2345 [2063 to 3006]
  Observed FTC-TP concentrations | 261 [152 to 341] | 976 [737 to 1359] | 4031 [2913 to 4342]

3. Primary Outcome: Concentrations of Tenofovir Disphosphate (TFV-DP) and Emtricitabine Triphosphate (FTC-TP) Measured at Four Weeks in Peripheral Blood Mononuclear Cells (PBMCs)
Description: Steady-state TFV-DP and FTC-TP concentrations observed in peripheral blood mononuclear cells (PBMCs) after ten weeks of directly observed therapy with TAF-FTC oral PrEP, in women randomized to receive 2, 4, or 7 doses per week, representing poor, moderate, or perfect adherence, respectively.
Time Frame: Assessed at week 4
Measure: Median (Inter-Quartile Range); unit: fmol/10^6 cells
Arm/Group | Poor Adherence | Moderate Adherence | Perfect Adherence
Number analyzed (Participants) | 17 | 17 | 18
fmol/10^6 cells
  Observed TFV-DP concentrations | 70 [55 to 94] | 229 [159 to 278] | 680 [462 to 864]
  Observed FTC-TP concentrations | 407 [337 to 500] | 1859 [1126 to 2990] | 6402 [4845 to 8010]

4. Primary Outcome: Fitted Steady-state TFV-DP Concentrations in Dried Blood Spots (DBS)
Description: Fitted steady-state TFV-DP concentrations after ten weeks of directly observed therapy with TAF-FTC oral PrEP, in women randomized to receive 2, 4, or 7 doses per week, representing poor, moderate, or perfect adherence, respectively.
Time Frame: Assessed through 10 weeks
Measure: Median (Inter-Quartile Range); unit: fmol/punch
Arm/Group | Poor Adherence | Moderate Adherence | Perfect Adherence
Number analyzed (Participants) | 18 | 18 | 18
fmol/punch | 468 [423 to 531] | 1010 [853 to 1231] | 2355 [1923 to 2609]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the ten weeks between randomization (i.e., administration of first dose of study product) and administration of the final dose of study product at the end of the directly observed therapy (DOT) phase.
Description: Adverse events meeting the following criteria were recorded: Clinical AEs of Grade 1 and above, laboratory AEs of Grade 2 and above, all AEs (clinical or laboratory) leading to a study product hold (temporary or permanent)
Groups:
- 2 doses per week (Poor Adherence): Cisgender women will receive a single tablet of coformulated 25 mg TAF/ 200mg FTC twice per week
- 4 doses per week (Moderate Adherence): Cisgender women will receive a single tablet of coformulated 25 mg TAF/ 200mg FTC 4 times per week
- 7 doses per week (Perfect Adherence): Cisgender women will receive a single tablet of coformulated 25 mg TAF/ 200mg FTC once daily (7 doses per week).
Arm/Group | 2 doses per week (Poor Adherence) | 4 doses per week (Moderate Adherence) | 7 doses per week (Perfect Adherence)
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 17/18 | 17/18 | 17/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 2 doses per week (Poor Adherence) (N=18) | 4 doses per week (Moderate Adherence) (N=18) | 7 doses per week (Perfect Adherence) (N=18)
Tonsilitis (Blood and lymphatic system disorders) | 1 | 1 | 2 — Grade 1 in all participants
Abdominal pain (Gastrointestinal disorders) | 3 | 2 | 1 — Grade 1 in all participants
Bloating (Gastrointestinal disorders) | 0 | 3 | 2 — Grade 1 in all participants
Gastritis (Gastrointestinal disorders) | 2 | 3 | 2 — Grade 1 in all participants
Vomiting (Gastrointestinal disorders) | 3 | 1 | 1 — Grade 1 in all participants
Nausea (Gastrointestinal disorders) | 8 | 7 | 6 — Grade 1 in all participants
Fatigue (General disorders) | 2 | 0 | 0 — Grade 1 in all participants
Flu-like symptoms (General disorders) | 0 | 2 | 0 — Grade 1 in all participants
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 2 — Grade 1 in all participants
Headache (Nervous system disorders) | 7 | 4 | 5 — Grade 1 in all participants
Urinary tract infection (Renal and urinary disorders) | 4 | 3 | 1 — Grade 1 in seven participants, Grade 2 in one participant
Breast pain (Reproductive system and breast disorders) | 1 | 0 | 2 — Grade 1 in all participants
Excessive spotting (Reproductive system and breast disorders) | 2 | 0 | 0 — Grade 1 in all participants
Pharyngitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 3 — Grade 1 in all participants
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 4 | 5 | 3 — Grade 1 in all participants
Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 7 — Grade 1 in all participants
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 3 | 3 — Grade 1 in all participants
Wound (Skin and subcutaneous tissue disorders) | 3 | 0 | 1 — Grade 1 in all participants
Fungal skin infection (Skin and subcutaneous tissue disorders) | 3 | 2 | 2 — Grade 1 in all participants

LIMITATIONS AND CAVEATS:
1. Dosing of TAF/FTC was up to only ten weeks.
2. Assessment of drug concentrations in PBMCs is highly dependent on cell processing and count protocols, meaning that it is difficult to compare PBMCs results across laboratories and studies.
3. The study did not explicitly evaluate the concentration-efficacy relationship.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2022-08-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT05140954/Prot_SAP_ICF_000.pdf